CLINICAL TRIAL: NCT00742755
Title: Increasing Adherence to Follow-up of Breast Abnormalities in Low-Income Korean American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: DAMD17-03-1-067
Record Dates: First submitted 2008-08-27; First posted 2008-08-28 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-02

CONDITIONS: Breast Cancer
Keywords: Follow-up of breast abnormalities; Korean American immigrants
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prospective Intervention (Experimental): Peer navigator intervention
  Interventions: Behavioral: Prospective intervention

INTERVENTIONS:
Behavioral: Prospective intervention — Prospective Intervention: Peer navigator who assists with appointment making, transportation, translations, completing forms, etc.
  Other Names: Intervention group

SUMMARY:
Develop and evaluate a peer navigator intervention to assist Korean women with a potential breast abnormality, who have missed their first follow-up appointment, to complete all diagnostic follow-up tests.

DETAILED DESCRIPTION:
The purpose of this study is to design an intervention to assist Korean American women who have been identified with a potential breast abnormality through the Breast Cancer Early Detection Program and who have missed their first follow-up appointment (at risk women). Intervention activities will include reminder phone calls or home visits by a trained peer navigator to explain the importance of follow-up procedures, emotional support, help with transportation to follow-up appointments, translations, organizing care for children or grandchildren during medical appointments, and other assistance to overcome barriers to follow-up identified during the initial phase of the study. The investigators will collect extensive process measures including number and type of intervention activities requested and delivered in order to estimate the feasibility for institutionalizing intervention activities. The investigators will conduct chart reviews and a follow-up survey to evaluate the effectiveness of the intervention in increasing adherence to follow-up procedures.

ELIGIBILITY:
Inclusion Criteria:

* Being: a Korean American woman
* Screened through the Breast Cancer Early Detection Program
* With a potential breast abnormality
* Having missed a first diagnostic follow-up appointment

Exclusion Criteria:

* Not a Korean American woman
* Not screened through the Breast Cancer Early Detection Program
* No potential breast abnormality
* Not having missed a first diagnostic follow-up appointment

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2003-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Completion of all recommended follow-up tests | 6 months post-intervention

SECONDARY OUTCOMES:
Time to completion | 6 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Annette E Maxwell, Dr.P.H., Principal Investigator — Division of Cancer Prevention and Control Research, University of California Los Angeles
Locations (1):
- Division of Cancer Prevention and Control Research, University of California Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Result] Maxwell AE, Jo AM, Crespi CM, Sudan M, Bastani R. Peer navigation improves diagnostic follow-up after breast cancer screening among Korean American women: results of a randomized trial. Cancer Causes Control. 2010 Nov;21(11):1931-40. doi: 10.1007/s10552-010-9621-7. Epub 2010 Jul 31. PMID 20676928